CLINICAL TRIAL: NCT06558253
Title: An Exploratory Study to Assess the Safety and Efficacy of Coenzyme I for Injection in Promoting Hematopoietic Recovery After Single-unit Unrelated Cord Blood Transplantation in Patients With Hematological Malignancies
Brief Title: The Safety and Efficacy of Coenzyme I for Injection in Promoting Hematopoietic Recovery of Patients After sUCBT
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: coenzyme I for injection
Record Dates: First submitted 2024-08-14; First posted 2024-08-16 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Hematopoietic Recovery
Keywords: Hematopoietic recovery, sUCBT
MeSH Terms: interventions — NAD; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Coenzyme I for Injection (Experimental): Subjects received 21 consecutive days of intravenous infusion of Coenzyme I for injection with three dose groups.
  Interventions: Drug: Coenzyme I for Injection

INTERVENTIONS:
Drug: Coenzyme I for Injection — Subjects received 21 consecutive days of intravenous infusion of Coenzyme I for injection, starting from the day of transplantation , and then continuously applied intravenously until 20 days post transplantation, with three dose groups: subjects #1-3 received one intravenous infusion per day containing 10 mg of Coenzyme I for injection, subjects #4-6 received one intravenous infusion per day containing 20 mg of Coenzyme I for injection, and subjects #7-12 received one intravenous infusion per day containing 50 mg of Coenzyme I for injection. Subjects in either dose group experienced a treatment-related Grade 3 or higher adverse reaction, the previous dose group was the maximum tolerated dose.

SUMMARY:
To assess the safety and efficacy of coenzyme I for injection in promoting hematopoietic recovery after single-unit unrelated cord blood transplantation in hematological malignancies.

DETAILED DESCRIPTION:
A single-center, open-label, dose-escalation study to assess the safety and efficacy of coenzyme I for injection in promoting hematopoietic recovery after single-unit unrelated cord blood transplantation in hematological malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years (inclusive) at screening; gender is not restricted;
* Diagnosed with hematological malignancies to receive sUCBT for the first time;
* No severe organ failure and no active infections
* ECOG performance status of 0-2;
* Voluntarily participating in the clinical trial, with full understanding of the trial details and having signed the informed consent form.

Exclusion Criteria:

* Those with severe organ dysfunction or disease, such as severe disease and dysfunction of the heart, liver, kidneys and pancreas;
* Pregnant patients;
* Patients and/or authorised family members who refuse to receive Coenzyme I for Injection;
* Any life-threatening disease, physical condition, or organ system dysfunction that, in the opinion of the investigator, may compromise patient safety and put the results of the study at undue risk; drug-dependent individuals; patients with uncontrolled psychiatric disorders; and individuals with cognitive impairment;
* Participants in other clinical studies affecting hematopoietic recovery within 3 months;
* Those who are considered by the investigator to be unsuitable for enrolment (e.g., those who anticipate that the patient will not be able to adhere to the examination and treatment due to financial or other issues).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-11-29 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Adverse Event(AE) | From the date of initial treatment to 30 days after transplantation
  Number of treatment-related adverse events as assessed by CTCAE v5.0

SECONDARY OUTCOMES:
Neutrophil engraftment time | 42 days post transplantation
  The first day of absolute neutrophil count ≥ 0.5×10^9/L for 3 consecutive days post transplantation.
Cumulative incidence of neutrophil engraftment on day 16 | 16 days post transplantation
  Cumulative incidence of neutrophil engraftment on day 16 post transplantation.
platelet engraftment time | 180 days post transplantation
  The first day of platelet count ≥ 20×10^9/L for 7 consecutive days without platelet transfusions for 7 consecutive days post transplantation.
Cumulative incidence of platelet engraftment on day 60 | 60 days post transplantation
  Cumulative incidence of platelet engraftment on day 60 post transplantation.
Cumulative incidence of primary graft failure on day 30 | 30 days post transplantation
  Cumulative incidence of primary graft failure on day 30 post transplantation.
Cumulative incidence of grade II-IV and III-IV acute GVHD on day 100 | 100 days post transplantation
  Cumulative incidence of grade II-IV and III-IV acute GVHD on day 100 post transplantation.
Cumulative incidence of transplant-related mortality on day 180 | 180 days post transplantation
  Cumulative incidence of transplant-related mortality on day 180 post transplantation.
Cumulative incidence of relapse on day 180 | 180 days post transplantation
  Cumulative incidence of relapse on day 180 post transplantation.
Probability of overall survival | 180 days post transplantation
  Probability of overall survival on day 180 post transplantation.
Probability of leukemia-free survival | 180 days post transplantation
  Probability of leukemia-free survival on day 180 post transplantation.
Probability of GVHD-free relapse-free survival | 180 days post transplantation
  Probability of GVHD-free relapse-free survival on day 180 post transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyu Zhu, Ph.D, Principal Investigator — The First Affiliated Hospital of University of Science and Technology of China
Locations (1):
- The First Affiliated Hospital of University of Science and Technology of China (Anhui Provincial Hospital), Hefei, Anhui, China